CLINICAL TRIAL: NCT00244530
Title: Postoperative Renal Function After Open-Heart Surgery in Patients With Impaired Renal Function Preoperatively. A Study of the Calcium Channel Blocker Nifedipine's Prophylactic Effect on Further Decline in Renal Function.
Brief Title: Prophylactic Effect of Nifedipine on Further Decline in Renal Function in Patients Undergoing Open-Heart Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oslo School of Pharmacy (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIF-123
Record Dates: First submitted 2005-10-25; First posted 2005-10-26 (Estimated); Last update posted 2006-12-22 (Estimated); Status verified 2006-12

CONDITIONS: Kidney Failure, Chronic; Coronary Artery Disease
Keywords: Preventive Therapy; Calcium Channel Blockers; Kidney Failure, Chronic; Coronary Artery Bypass; Heart Valve Prosthesis Implantation
MeSH Terms: conditions — Kidney Failure, Chronic; Coronary Artery Disease | interventions — Nifedipine

INTERVENTIONS:
Drug: Nifedipine

SUMMARY:
To compare renal function (51Cr-EDTA clearance) 48 hours post open-heart surgery (coronary bypass or valve surgery) in patients with impaired renal function after randomization to either nifedipine infusion at start of surgery and the following 24 hours or placebo (0.9% saline infusion). Study hypothesis is that nifedipine has a prophylactic effect on decline in renal function.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either gender above 18 years of age.
2. Patients with significant coronary stenosi(e)s (≥ 75% coronary artery lumen surface stenosi(e)s and / or aortic- or mitral valve vitriuim that are accepted for coronary artery bypass surgery and/or valve replacement surgery.
3. Patients with impaired renal function, defined as increased serum- creatinine. Men: ≥ 150 µmol/l and Women: ≥130 µmol/l.

Exclusion Criteria:

1. Patients on maintenance hemodialysis
2. Renal transplant patients
3. Patients with ejection fraction ≤ 35%
4. Patients with unstable angina pectoris

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2001-06; Study Completion 2005-10

PRIMARY OUTCOMES:
Primary efficacy endpoint is change in renal function, evaluated by 51Cr-EDTA clearance between 24 hours pre open-heart surgery and 48 hours post open-heart surgery. Sample size is 20, ten in each group.

SECONDARY OUTCOMES:
Change in renal function after open-heart surgery, as measured by cimetidine refined serum creatinine clearance with measurements preoperatively and 2-6 hours, 20-24 hours and 44-48 hours postoperatively. Need for dialysis post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Jan F Bugge, MD, PhD, Study Chair — Rikshospitalet University Hospital, Oslo, Norway
Locations (1):
- Rikshospitalet University Hospital, Oslo, Norway